CLINICAL TRIAL: NCT00793663
Title: 1) The Effect of Xenon and Sevoflurane on Hypnosis Monitors. 2) Prevention of Postoperative Nausea and Vomiting. 3) Rescue Treatment of Established Postoperative Nausea and Vomiting. Sevoflurane.
Brief Title: Depth of Hypnosis and Postoperative Nausea and Vomiting During Xenon Anaesthesia
Acronym: XABP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Air Liquide Santé International (Industry)
Responsible Party: Dr Mark Coburn, Principal Investigator, RWTH Aachen University; Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALS-8-08-A-401; EudraCT-number:; 2008-004132-20; Protocol version:; Version V3; Date: 20.10.2008
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Anaesthetics Gases, Xenon; Anaesthetics Volatile, Sevoflurane; Depth of Anaesthesia; Postoperative Nausea; Postoperative Vomiting
Keywords: Xenon; Sevoflurane; Postoperative Nausea and vomiting; Depth of anaesthesia
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Xenon; Sevoflurane; Dexamethasone; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): The effect of xenon as an anaesthetic on the depth of hypnosis.
  Interventions: Drug: Xenon
- 2 (Active Comparator): The effect of sevoflurane as an anesthetic on the depth of hypnosis
  Interventions: Drug: Sevoflurane
- 3 (Experimental): Dexamethasone as prevention of postoperative nausea and vomiting after xenon or sevoflurane anesthesia
  Interventions: Drug: Dexamethasone
- 4 (Placebo Comparator)
  Interventions: Drug: NaCl
- 5 (Experimental): Ondansetron, to determine the onset-time of ondansetron when used as rescue medication for postoperative nausea and vomiting
  Interventions: Drug: Ondansetron
- 6 (Placebo Comparator)
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: Xenon — Inhalational gas; maximum dose allowed: 70 % Xenon; the duration of the treatment will be defined through anesthesia-time.
  Other Names: LENOXe
  Arms: 1
Drug: Sevoflurane — Inhalation gas; age adapted MAC-values; the duration of the treatment will be defined through anesthesia-time
  Other Names: Sevorane
  Arms: 2
Drug: Dexamethasone — Intravenous use, 4 mg, single shot
  Other Names: Fortecortin Inject
  Arms: 3
Drug: NaCl — Intravenous use; single shot
  Arms: 4
Drug: Ondansetron — Intravenous use; 4 mg; single shot
  Other Names: Zofran
  Arms: 5
Drug: NaCl — Intravenous use; single shot
  Arms: 6

SUMMARY:
The purpose of this study is ad 1) to measure the depth of hypnosis as assessed by BIS and cAAI during an average general anesthesia with xenon or sevoflurane and to establish a reliable monitoring system for measuring and documenting the actual depth of hypnosis for the volatile anesthetics investigated. Ad 2) the question is to be answered whether 4 mg dexamethasone i.v. is an effective prophylactic treatment against postoperative nausea and vomiting in case of xenon or sevoflurane anesthesia. Ad 3) it serves to gain evidence about the (non-)effectiveness and kinetics of ondansetron as antiemetic remedy after xenon or sevoflurane anesthesia.

DETAILED DESCRIPTION:
1. Patients included into the trial will randomly be allocated to either 0.8-1.1 minimum alveolar concentration (MAC) xenon in 30 % oxygen or 0.8-1.1 MAC sevoflurane (age adapted)/30 % oxygen. The MAC is defined and will therefore be applied according to the investigated subject's age. Premedication will be performed with midazolam 7.5 mg orally 45 min before induction (standard dose and application form for adults as clinical practice of our department). Anesthesia will be induced in both groups with propofol 2 mg/kg i.v. and remifentanil 0.5 mcg/kg/min by infusion over 60 s. For tracheal intubation non-depolarizing neuromuscular blocking agents can be used (rocuronium 0.6 mg/kg). Both groups will receive remifentanil at a base rate of 0.2 mcg/kg/min. Xenon or sevoflurane can be titrated in the range from 0.8-1.1 MAC according to clinical needs based on the patient's hemodynamic, autonomic and somatic signs. Twenty minutes before the estimated cessation of all surgical procedures 0.05 mg kg-1 piritramide for post anesthetic pain management will be administered intravenously, as well as a short infusion of metamizole 15 mg kg-1.

   Depth of anesthesia (hypnosis) will be monitored with spontaneous EEG (BIS VISTA, Aspect Medical Systems, Newton, MA) and the mid latency auditory evoked potentials including a monitoring variable indicating the patients hypnotic state calculated from the MLAEP and the electroencephalogram, the composite A-Line ARX Index (cAAI) with the AEP Monitor/2 (Danmeter A/S, Odense, Denmark). Dosing will be conducted according to the current clinical standard without the monitoring, thus the anesthesia provider will be blinded towards both measurements.
2. After induction of anesthesia patients will be randomized to a second factor, i.e. 4 mg dexamethasone or placebo for the prevention of PONV. To avoid potential imbalances, this will be achieved using a factorial design. The application of dexamethasone or placebo will be blinded to the investigator assessing postoperative nausea and vomiting.
3. Patients who experience significant nausea will be randomized to receive either 4 mg ondansetron or placebo and the course of nausea will be assessed for > 32 min. Again, the application of ondansetron or placebo will be blinded to the investigator assessing postoperative nausea and vomiting. If the symptoms of postoperative nausea and vomiting persist for more than 32 min after treatment additional rescue treatment will be offered. Of note, all patients are able to receive further rescue treatment at any time point of the study on demand.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 < 75 years
* ASA physical status I-II
* planned duration of anesthesia ≥ 60 minutes
* Apfel score ≥ 2-3
* elective (laparoscopic) surgery (abdominal, gynecological)
* women: with a highly effective contraception, defined as methods with a pearl index < 1 (i.e. hormonal contraceptives, IUD)

Exclusion Criteria:

* history of hypersensitivity to any used drugs or additive components used for preparation and stabilization of the named drugs in this trial
* history or reasonable suspicion of malignant hyperthermia and/or degenerative neuromuscular disease, in the subject observed or blood relatives
* history of liver function disorders, leucocytosis and unclear fever after usage of halogenated anesthetics.
* any indisposition that may be aggravated by the use of the drugs investigated:
* liver and/or kidney function disorders
* severe acute or chronic infectious disease (i.e. viral, bacterial, fungal)
* elevated intracranial pressure
* history of gastrointestinal ulcer(s) or inflammatory bowel disease
* severe metabolic disorders
* hematoporphyria
* glaucoma
* hearing disorders
* any disease including air-filled closed cavities, such as pneumothorax, ileus
* pregnancy and lactation period
* subjects under the age of 18 years
* ambulatory surgery
* any disease that is associated with the requirement of a high oxygen yield and/or
* risk of high oxygen consumption:
* severe lung and/or airway disease
* coronary heart disease and/or seriously impaired cardiac function
* severe psychiatric disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The average depths of hypnosis as assessed by the BIS and the cAAI between skin incision and start of closure. | During anaesthesia
Postoperative nausea as assessed by a verbal rating scale (VRS) ranging between 0 and 10. | After anesthesia at 5, 10, 15, 30, 45, 60, and 90 min. At 2, 6 and 24 h after anesthesia the maximum nausea will be rated for the 30-120 min, 2-6 h, and 6-24 h interval.
Reduction of VRS nausea immediately at 2, 5, 7.5, 10, 15, 20 and 30 min after rescue treatment administration. | Maximum nausea will be rated at 2, 6 and 24 hours after treatment for the 30-120 min, 2-6 h and 6-24 h interval.

SECONDARY OUTCOMES:
Heart rate and blood pressure | During anesthesia
Observer´s assessment of alertness and sedation scales | Recovery from anesthesia
Sensitivity and specificity characteristics for both the BIS and the cAAI. | During anesthesia
Awareness after anesthesia assessed by the Brice questionnaire at 2 and 24 hours after anesthesia. | 24 hours after anaesthesia
Occurrence of postoperative vomiting and the respective time-points will be recorded. Postoperative vomiting is defined as vomiting or retching. | 24 hours postoperative
Usage of rescue medication, time and dosage | 24 hours postoperative
Time to discharge from post anesthetic care unit (Aldrete Score ≥ 9 equals the hypothetic discharge time from post anesthetic care unit) | Time in the post anesthetic care unit

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Rossaint, MD, Study Chair — RWTH University Aachen; Department of Anesthesiology
Locations (1):
- RWTH Aachen University; Department of Anesthesiology, Aachen, Germany

REFERENCES:
- [Derived] Fahlenkamp AV, Stoppe C, Cremer J, Biener IA, Peters D, Leuchter R, Eisert A, Apfel CC, Rossaint R, Coburn M. Nausea and Vomiting following Balanced Xenon Anesthesia Compared to Sevoflurane: A Post-Hoc Explorative Analysis of a Randomized Controlled Trial. PLoS One. 2016 Apr 25;11(4):e0153807. doi: 10.1371/journal.pone.0153807. eCollection 2016. PMID 27111335